CLINICAL TRIAL: NCT01414478
Title: A Prospective, Randomized Trial to Evaluate the Efficacy of High Protein Intake on the Incidence of Emesis and Promotion of Patient Satisfaction After Epidural Analgesia for Labor
Brief Title: High Protein Intake to Decrease Emesis and Promote Patient Satisfaction in Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO10070074
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-02

CONDITIONS: Emesis
Keywords: emesis; nausea
MeSH Terms: conditions — Vomiting; Nausea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Protein Shake (Active Comparator): Protein shake that contain 30 grams of protein in 11 fluid ounces.
  Interventions: Other: Protein Shake
- Ice Chips (No Intervention): Patients allowed consumption of ice chips only during labor.

INTERVENTIONS:
Other: Protein Shake — Protein shake contains 30 grams of protein in 11 fluid ounces.
  Other Names: Premier Nutrition Protein Shake
  Arms: High Protein Shake

SUMMARY:
The purpose of our study is to determine if the incidence of emesis can be lowered with the addition of a high protein drink during labor. Emesis and nausea are the leading causes of parturient dissatisfaction, results in a delay of returning to normal, daily living and can hugely impact the mother's postpartum experience. To date, no studies have been done on the relationship of protein intake during labor and incidence of emesis. To the best of our knowledge, the use of a high protein drink during labor has not been evaluated in the literature.

DETAILED DESCRIPTION:
The investigators plan to enroll women (n=150) who requested epidural anesthesia for labor. After placement of their labor epidural catheter, parturients will be randomized by a computer generated number table into one of two groups. Group P - high protein drink with 30 grams of protein and ice chips PRN, or Group C - control group consisting of ice chips PRN. The protein drink that will be used is Premier Nutrition Protein Shake, which contains 30 grams of protein in 11 ounces. Measured variables will include; nausea and emesis at epidural placement, at hourly intervals until delivery, and 1 hour post delivery. Nausea will be evaluated using a visual analog scale (VAS); 0 = no nausea and 10 = worst nausea ever. Episodes of emesis will be recorded as (yes/no). The parturient will be seen the day following delivery and evaluated for overall patient satisfaction. Parturients will rate their satisfaction level using a scale from 0-100 with 0=not satisfied and 100=very satisfied. The investigators believe that the incidence of emesis will be decreased in parturients who receive high protein intake during labor, and overall patient satisfaction will be increased.

ELIGIBILITY:
Inclusion Criteria:

All women of childbearing age who request labor epidural analgesia, ≤ 5cm cervical dilatation at the time of epidural insertion, > 36 weeks gestation, singleton pregnancy, vertex presentation, and NPO more than 4 hours prior to epidural insertion. Both nulliparous and multiparous women will be included. Minors under the age of 18 years will be included and a separate informed consent will be presented to these individuals.

Exclusion Criteria:

Women with diabetes (at increased risk for gastroparesis and fetal macrosomia), multiple gestation, non-vertex fetal presentation, chronic opioid use (delayed gastric emptying), history of gastric bypass surgery (abnormal anatomical stomach), severe morbid obesity (BMI > 40kg/m2 due to increased intragastric pressure), and history of known obstetric or medical complication (i.e. preeclampsia) that may increase the likelihood of a complicated or operative delivery (i.e. cesarean section).

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2010-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Emesis in labor | Throughout labor (up to one hour post delivery)
  To determine the incidence of emesis after high protein intake in parturients who have received labor epidural analgesia up until one hour post delivery.

SECONDARY OUTCOMES:
Patient satisfaction with labor after consumption of a high protein shake. | Throughout labor (up to 24 hours post delivery)
  Our secondary aim is to determine the incidence of nausea after high protein intake during labor and overall parturient satisfaction with their birthing experience 24 hours post delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel C Vallejo, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital Women Care Birth Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Vallejo MC, Cobb BT, Steen TL, Singh S, Phelps AL. Maternal outcomes in women supplemented with a high-protein drink in labour. Aust N Z J Obstet Gynaecol. 2013 Aug;53(4):369-74. doi: 10.1111/ajo.12079. Epub 2013 Apr 4. PMID 23551108